CLINICAL TRIAL: NCT03891823
Title: EValuation of Outcomes of MitraCLip for the Treatment of Moderate Functional Mitral ValvE Regurgitation In Heart Failure
Brief Title: Transcatheter Mitral Valve Repair for the Treatment of Mitral Valve Regurgitation In Heart Failure (The EVOLVE-MR Trial)
Acronym: EVOLVE-MR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Montreal Heart Institute (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHICC-2018-002
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Ventricular Remodeling, Left
MeSH Terms: conditions — Ventricular Remodeling | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Randomized study of MitraClip vs. medical therapy in symptomatic heart failure patients with moderate (2+, 2-3+) functional mitral regurgitation and left ventricular dysfunction.
  Subjects will be followed for 24 months and there will be one formal interim analysis for futility after approximately 50% of subjects have completed their 24-month follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitraClip (Experimental): Study of MitraClip in symptomatic heart failure patients with moderate (2+, 2-3+) functional mitral regurgitation and left ventricular dysfunction.
  Subjects will be followed for 24 months and there will be one formal interim analysis for futility after approximately 50% of subjects have completed their 24-month follow-up.
  Interventions: Device: MitraClip; Drug: Medical Therapy
- Medical Therapy (Active Comparator): Study of medical therapy in symptomatic heart failure patients with moderate (2+, 2-3+) functional mitral regurgitation and left ventricular dysfunction.
  Subjects will be followed for 24 months and there will be one formal interim analysis for futility after approximately 50% of subjects have completed their 24-month follow-up.
  Interventions: Device: MitraClip; Drug: Medical Therapy

INTERVENTIONS:
Device: MitraClip — Study participants will be randomized to MitraClip device to determine treatment efficacy in improving LV remodelling or functional capacity.
Drug: Medical Therapy — Study participants will be randomized to medical therapy to determine treatment efficacy in improving LV remodelling or functional capacity.

SUMMARY:
The study compares the effectiveness of treatment with MitraClip to medical therapy in improving the reduction of cardiovascular morbidity and functional capacity at 24 months, in patients with moderate functional mitral regurgitation.

DETAILED DESCRIPTION:
Primary Objective To compare the effectiveness of treatment with MitraClip to medical therapy on the change from baseline to 24 months in quality of life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score in patients with moderate functional mitral regurgitation.

Secondary Objectives

* To evaluate the effects of MitraClip and medical therapy on change from baseline in mitral regurgitation severity at 24 months.
* To evaluate the effects of MitraClip and medical therapy on change from baseline in mitral regurgitation severity at 12 months.
* To evaluate the effects of MitraClip and medical therapy on change in quality of life from baseline to 12 months, as measured by the KCCQ.

Tertiary Objectives

* To evaluate the effects of MitraClip and medical therapy on change from baseline in functional capacity (distance walked on a 6MWT) at 12 and 24 Months.
* To evaluate the effects of MitraClip and medical therapy on change from baseline in quality of life, as measured by the EQ5DL questionnaire, at 12 and 24 months.
* To evaluate the effects of MitraClip and medical therapy on freedom from progression to severe MR at 24 months as assessed by echocardiography.
* To evaluate the effects of MitraClip and medical therapy on change from baseline in LVEDVi at 24 months.

Exploratory Objectives

* To evaluate the effects of MitraClip and medical therapy on functional class, biomarkers, clinical events, parameters of physical activity, other echocardiographic parameters and health economic assessments.
* To evaluate the effects of MitraClip and medical therapy on all hospitalizations for decompensated heart failure, including episodes of outpatient treatment intensification in a HF clinic or emergency department visits, at 24 months.

ELIGIBILITY:
Inclusion Criteria

Study participants must meet ALL of the following inclusion criteria in order to be eligible for this study:

1. Male or female ≥18 years of age;
2. Moderate (2+,2-3+) functional mitral regurgitation due to cardiomyopathy of either ischemic or non-ischemic etiology as determined by transthoracic echocardiogram (TTE), and confirmed by the Echocardiography Core Lab (ECL);
3. Left ventricular ejection fraction (LVEF) >20%, as determined by transthoracic echocardiogram (TTE), and confirmed by the Echocardiography Core Lab (ECL);
4. Symptomatic heart failure as defined by NYHA class II, III or ambulatory IV and NT-proBNP as follows:

   * NT-proBNP > 300 pg/mL in patients with sinus rhythm
   * NT-proBNP > 600 pg/mL in patients with atrial fibrillation
5. Treatment and compliance with medical therapy for heart failure for at least 30 days;

   Optimal medical therapy is defined by:

   a. Maximum tolerated beta-blocker, angiotensin converting enzyme inhibitor (ACE) or angiotensin receptor blocker (ARB), Entresto (valsartan/sacubitril), Ivabradine and aldosterone antagonist (as per the ACC/AHA Guidelines and Canadian Cardiovascular Society Heart Failure Guidelines or other therapies (including SGLT2 inhibitors) as judged by the HF specialist investigator on site and confirmed by the Clinical Eligibility Committee.
6. Clinical agreement amongst local investigators that the patient will not be offered surgical intervention;
7. The primary regurgitant jet, in the opinion of the MitraClip implanting investigator, can successfully be treated by the MitraClip. Treatment of commissural mitral regurgitation may be treated at the discretion of the operator. All major jets contributing the secondary MR will be treated with the MitraClip;
8. Ability to perform a six-minute walk test (6MWT) without substantial physical limitations and without use of a walker or wheelchair and distance walked in 6 minutes of ≤ 450m;
9. Ability and willingness to give written informed consent and to comply with the requirements of the study.

Exclusion Criteria

Study participants meeting any of the following exclusion criteria by the day of randomization (visit 1) are NOT eligible for this study:

1. Life expectancy less than 12 months due to non-cardiac conditions;
2. ACC/AHA Stage D Heart Failure;
3. Left ventricular ejection fraction ≤ 25%; indexed left ventricular end-diastolic volume ≥100 ml/m2;
4. Severe (3-4+, 4+) secondary mitral regurgitation with an indication for intervention;
5. Hypotension (systolic pressure <90 mm Hg) or requirement for inotropic support or mechanical hemodynamic support;
6. United Network for Organ Sharing (UNOS) status 1 heart transplantation (Canadian Cardiac Transplantation Network, CCTN, status 4) or prior orthotopic heart transplantation;
7. Untreated clinically significant coronary artery disease requiring revascularization;
8. CABG within prior 30 days;
9. Percutaneous coronary intervention within prior 30 days;
10. Severe Chronic Obstructive Pulmonary Disease (COPD) requiring continuous daytime home oxygen or chronic oral corticosteroid therapy;
11. Previous surgical mitral valve bioprosthesis, mitral annuloplasty, or transcatheter mitral valve procedure;
12. Positive pregnancy test, or woman of child bearing potential not using highly effective methods of contraception;

    Women are considered not of childbearing potential if they:
    1. Have had a hysterectomy, a bilateral oophorectomy or tubal ligation prior to Baseline Visit.
    2. Are postmenopausal defined as no menses for at least 1 year and have a serum FSH level of 40 IU/L.

    Women of childbearing potential must agree to use an effective method of birth control throughout the study. Acceptable means of birth control include: implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, male or female condoms with spermicide, abstinence, or a sterile sexual partner.
13. Mitral valve area <4.0 cm2 as assessed by planimetry of the mitral valve;
14. Subjects in whom trans-esophageal echocardiography is contraindicated or is at high risk;
15. Mitral leaflet anatomy which may preclude MitraClip implantation:

    1. Perforated mitral leaflets or clefts, lack of primary or secondary chordal support;
    2. Severe calcification in the grasping area;
    3. Rheumatic valve disease.
16. Stroke or transient ischemic event within 30 days before randomization;
17. Modified Rankin Scale >4 disability;
18. Need for emergent or urgent surgery for any reason or any planned cardiac surgery within the next 12 months;
19. Severe renal impairment defined as an Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73m2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula;
20. Severe anemia requiring transfusional support or therapy with erythropoietin;
21. Physical evidence of uncontrolled right-sided congestive heart failure with echocardiographic evidence of moderate or severe right ventricular dysfunction;
22. Aortic valve disease requiring surgery or transcatheter intervention;
23. Significant tricuspid valve disease requiring surgical intervention or very severe tricuspid regurgitation with evidence of right ventricular dysfunction;
24. Active infection requiring antibiotic therapy;
25. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease;
26. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
27. Any condition making it unlikely the patient will be able to complete all protocol procedures (including compliance with guideline-directed medical therapy) and follow-up visits;
28. Presence of any of the following:

    1. Pulmonary artery systolic pressure (PASP) > 70 mm Hg confirmed by right heart catheterization;
    2. Infiltrative cardiomyopathies.
29. Any other condition(s) that would compromise the safety of the patient as judged by the site principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Change In Mitral Regurgitation | 24 months
  To compare the effectiveness of treatment with MitraClip to medical therapy on the change from baseline to 24 months in quality of life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score in patients with moderate functional mitral regurgitation

SECONDARY OUTCOMES:
Change in Mitral Regurgitation Severity at 24 Months | 24 months
  To evaluate the effects of MitraClip and medical therapy on change from baseline in mitral regurgitation severity at 24 months.
Change in Mitral Regurgitation Severity at 12 Months | 12 months
  To evaluate the effects of MitraClip and medical therapy on change from baseline in mitral regurgitation severity at 12 months.
Change in Quality of Life Assessment | 12 months
  To evaluate the effects of MitraClip and medical therapy on change in quality of life from baseline to 12 months, as measured by the KCCQ.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Rouleau, MD, Principal Investigator — Montreal Heart Institute; Anique Ducharme, MD, Principal Investigator — Montreal Heart Institute; Sophie Tanguay, MSc, Study Director — Montreal Health Innovations Coordinating Centre
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No